CLINICAL TRIAL: NCT04347863
Title: Investigating Program of Food Preparation on Diet Improvement for Patients With Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taiwan Adventist Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 106-E-29
Record Dates: First submitted 2020-04-13; First posted 2020-04-15 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Stroke; Dysphagia, Late Effect of Stroke
Keywords: Food preparation; Dietary well-being; Quality of life; Dysphagia; Stroke
MeSH Terms: conditions — Stroke; Deglutition Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Group swallowing disorder diet preparation program
  Interventions: Other: Group swallowing disorder diet preparation program
- Control group (No Intervention): No Intervention

INTERVENTIONS:
Other: Group swallowing disorder diet preparation program — This program included food properties, select food, type of cooking, using thickener and tasting
  Arms: Experimental group

SUMMARY:
This is a randomized controlled behavioral intervention trial to assess the efficacy of investigating program of food preparation on diet improve patients with stroke.

DETAILED DESCRIPTION:
This is a randomized controlled behavioral intervention trial to assess the efficacy of investigating program of food preparation on diet improve patients with stroke. Subjects will be randomized to intervention group and control group.The primary outcome included seven measures, Functional oral intake scale, Mini Nutritional Assessment, Council on Nutrition Appetite Questionnaire, Dietary Well-Being Scale, Swallowing Quality of Life questionnaire, WHO Quality of Life-BREF and Eating Assessment Tool-10.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis is stroke
* EAT-10 ≥ 3
* Aged > 20 years
* Capability of following instructions
* Willing to participants to the study

Exclusion Criteria:

* Non-stroke neurological diseases ( ex: traumatic brain injury, brain tumor, neurodegenerative disease and Parkinson's disease )
* Dysphagia by neck injury or surgery
* During the study, he/she was hospitalized again due to disease.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-04-19 (Actual); Primary Completion 2018-09-28 (Actual); Study Completion 2018-09-28 (Actual)

PRIMARY OUTCOMES:
Changes of the Eating Assessment Tool-10 | 6 weeks
  Eating Assessment Tool-10 assesses ability of swallowing by myself. The total scare ranges from 0-40. A higher level indicates better ability of swallowing. Changes of the Eating Assessment Tool-10 will be assessed before and after intervention.
Changes of the Functional Oral Intake Scale | 6 weeks
  Functional Oral Intake Scale assesses ability of swallowing. The total level ranges from 1-7. A higher level indicates better ability of swallowing. Changes of the Functional Oral Intake Scale will be assessed before and after intervention.
Changes of the Mini Nutritional Assessment | 6 weeks
  Mini Nutritional Assessment assesses comprehensive nutritional. The total score ranges from 0-30. A higher score indicates better nutrition status. Changes of the Mini Nutritional Assessment will be assessed before and after intervention.
Changes of the Council on Nutrition Appetite Questionnaire | 6 weeks
  Council on Nutrition Appetite Questionnaire assesses appetite.The total score ranges from 8-40. A higher score indicates better appetite. Changes of the Council on Nutrition Appetite Questionnaire will be assessed before and after intervention.
Changes of the Dietary Well-Being Scale | 6 weeks
  Dietary Well-Being Scale assesses dietary well-being. The total scare ranges from 21-126. A higher score indicates better dietary well-being. Changes of the Dietary Well-Being Scale well be assessed before and after intervention.
Changes of the Swallowing Quality of Life questionnaire | 6 weeks
  Swallowing Quality of Life questionnaire assesses quality of life about swallowing.The total score ranges from 44-220. A higher score indicates better quality of life about swallowing. Changes of the Swallowing Quality of Life questionnaire well be assessed before and after intervention.
Changes of the WHO Quality of Life-BREF | 6 weeks
  WHO Quality of Life-BREF assesses quality of life. The total score ranges from 28-140. A higher score indicates better quality of life. Changes of the WHO Quality of Life-BREF well be assessed before and after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: En-Chi Chiu, PhD, Study Director — National Taipei University of Nursing and Health Sciences
Locations (1):
- National Taipei University of Nursing and Health Sciences, Taipei, Beitou Dist, Taiwan